CLINICAL TRIAL: NCT05541055
Title: Clinical Effectiveness of Digital CBT-I for the Treatment of Insomnia Disorder: A Randomized Controlled Trial
Brief Title: Digital CBT-I for Insomnia Disorder
Acronym: CrEDIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Big Health Inc. (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BH-S-01
Record Dates: First submitted 2022-09-07; First posted 2022-09-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Insomnia Disorder
Keywords: Insomnia; digital CBT; CBT-I
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Digital CBT-I (Experimental): Digitally-delivered CBT for insomnia accessed via web and/or mobile app
  Interventions: Device: digital CBT-I
- Sleep hygiene education (Active Comparator): This group will receive access to sleep hygiene education delivered via digital written materials
  Interventions: Other: Sleep hygiene education

INTERVENTIONS:
Device: digital CBT-I — A fully-automated and personalized digital intervention based on principles from cognitive behavioral therapy for insomnia.
  Other Names: Sleepio
  Arms: Digital CBT-I
Other: Sleep hygiene education — Participants will be provided with sleep hygiene advice which will be delivered digitally all at once upon allocation to the SHE arm. Participants will be able to revisit content during the trial as they wish.
  Arms: Sleep hygiene education

SUMMARY:
This study will examine the effectiveness of digital CBT-I versus sleep hygiene education in reducing insomnia severity, sleep onset latency, and wake after sleep onset in those with insomnia disorder.

DETAILED DESCRIPTION:
This study aims to examine the effectiveness of a fully-automated web and app-based digital CBT-I for insomnia compared to sleep hygiene education (SHE) in individuals with a diagnosis of insomnia disorder. Primary outcomes of interest include changes in insomnia severity, sleep onset latency, and wake after sleep onset throughout the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥22 years old
* Insomnia Disorder diagnosis
* Score ≤16 on the 8-item Sleep Condition Indicator
* > 30 minutes sleep onset latency (SOL); and/or > 30 minutes wake after sleep onset (WASO)
* Current resident of the USA
* Oral and written fluency in English
* Participant is able and willing to comply with protocol requirements, has been informed of the nature of the study, and has signed the IRB-approved informed consent form

Exclusion Criteria:

* Must not be currently receiving or be expecting to start CBT for insomnia during study participation, or have previously received CBT for insomnia in the past 12-months (self-report)
* If on psychoactive medication, including sleep medication, this must be stable for at least 5 half lives
* Past or present psychosis, schizophrenia, bipolar disorder, assessed by self-report and/or seizure disorder
* Occupation that requires alertness / caution to avoid accidents, for example long-haul driving, long distance bus driver, heavy machinery operator, air traffic controller
* Hearing or vision impairment that prevents effective use of the audio-visual content of digital CBT-I or SHE in the opinion of the investigator
* Intellectual disability or any Neurocognitive or Neurodevelopmental disorder that would prevent participants from following study procedures
* Any condition that the investigator believes would make participation in the study not in the best interest of the participant or would preclude successful completion of study activities

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Change in the Insomnia Severity Index (ISI) | From baseline to 10 weeks post-randomization
  Validated questionnaire; a 7-item scale with total scores between 0 and 28 where higher scores indicate greater severity
Change in sleep onset latency (SOL) | From baseline to 10 weeks post-randomization
  Measured by daily sleep diaries (based on the Consensus Sleep Diary) averaged across 10 days
Change in wake after sleep onset (WASO) | From baseline to 10 weeks post-randomization
  Measured by daily sleep diaries (based on the Consensus Sleep Diary) averaged across 10 days

SECONDARY OUTCOMES:
Insomnia Disorder remission (score <8) and response (change ≥6) on the ISI | 10, 16, and 24 weeks post-randomization
  Validated questionnaire; a 7-item scale with total scores between 0 and 28 where higher scores indicate greater severity
Insomnia disorder remission based on the SCID Insomnia Module | Week -1 compared to weeks 10, 16, and 24 post-randomization
  structured interview to assess for Insomnia Disorder
Change in sleep diary parameters: percent sleep efficiency (SE), total sleep time (TST), total time in bed (TTIB), and total wake time (TWT) | From lead-in period to 10, 16, and 24 weeks post-randomization
  Each measured in minutes by daily sleep diaries (based on the Consensus Sleep Diary)
Change in the Sleep Condition Indicator (SCI-8) | From baseline to weeks 10, 16, and 24 post-randomization
  Validated questionnaire; an 8-item scale with total scores between 0 and 32 where higher scores indicate better sleep
Change in the Generalized Anxiety Disorder Questionnaire (GAD-7) | From baseline to weeks 10, 16, and 24 post-randomization
  Validated questionnaire; a 7-item scale with total scores between 0 and 21 where higher scores indicate greater severity
Change in the Patient Health Questionnaire (PHQ-8) | From baseline to weeks 10, 16 and 24 post-randomization
  Validated questionnaire; an 8-item scale with total scores between 0 and 24 where higher scores indicate greater severity
Change in the Insomnia Severity Index (ISI) | From baseline to weeks 16 and 24 post-randomization
  Validated questionnaire; a 7-item scale with total scores between 0 and 28 where higher scores indicate greater severity
Change in sleep onset latency (SOL) | From baseline to weeks 16 and 24 post-randomization
  Measured by daily sleep diaries (based on the Consensus Sleep Diary) averaged across 10 days
Change in wake after sleep onset (WASO) | From baseline to weeks 16 and 24 post-randomization
  Measured by daily sleep diaries (based on the Consensus Sleep Diary) averaged across 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prather AA, Krystal AD, Emsley R, Carl J, Ball T, Tarnai K, Aguilera A, Espie CA, Henry AL. The Effectiveness of Digital Cognitive Behavioral Therapy to Treat Insomnia Disorder in US Adults: Nationwide Decentralized Randomized Controlled Trial. JMIR Ment Health. 2025 Dec 4;12:e84323. doi: 10.2196/84323. PMID 41343796